CLINICAL TRIAL: NCT05979896
Title: A Study Protocol to Assess the Chemoprevention Efficacy of Sulphadoxine-Pyrimethamine Plus Amodiaquine (SPAQ) and Resistance Marker Prevalence in Children 3-59 Months in Sokoto and Kwara States, Nigeria.
Brief Title: Chemoprevention Efficacy Study Nigeria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malaria Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SMCNGPHASE1
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Malaria
Keywords: Seasonal Malaria Chemoprevention; Chemoprevention efficacy; Antimalarial drug resistance
MeSH Terms: conditions — Malaria | interventions — Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sulfadoxine-Pyrimethamine + Amodiaquine (SPAQ) (Experimental): Children aged 3-59 months will receive directly observed therapy of standard aged based dosing of Sulfadoxine-Pyrimethamine + Amodiaquine (SPAQ) over 3 days.
  Interventions: Drug: Standard age based SPAQ administration for SMC

INTERVENTIONS:
Drug: Standard age based SPAQ administration for SMC — Sulfadoxine-pyrimethamine and amodiaquine (SPAQ) is administered in standard WHO approved age based regimens as used in Seasonal Malaria Chemoprevention Programmes.
  Sulphadoxine is a slowly eliminated sulphonamide. It is used in a fixed dose combination of 20 parts sulphadoxine with 1 part pyrimethamine given orally or intramuscularly.
  Sulphadoxine is readily absorbed from the GIT. It is widely distributed in body tissues and fluids and crosses the placenta into foetal circulation. It is also readily detectable in breast milk. It is excreted predominantly as the unchanged drug. AQ Amodiaquine is a Mannich base 4 amino-quinoline that interferes with parasite haem detoxification. It is more effective than chloroquine in both chloroquine sensitive and resistant P. falciparum infections. However, there is cross-resistance between chloroquine and amodiaquine.
  It is readily absorbed in the GIT and rapidly converted in the liver to the active metabolite, desethylamodiaquine.

SUMMARY:
The study aims to assess the chemoprevention efficacy of Sulfadoxine-Pyrimethamine and Amodiaquine (SPAQ) used in standard age-based dosing regimens used in Seasonal Malaria Chemoprevention (SMC) and SPAQ resistance marker prevalences and assocations among children 3 - 59 months in Sokoto and Kwara States, Nigeria.

DETAILED DESCRIPTION:
The study aims (1) to determine the chemoprevention efficacy of Sulfadoxine-Pyrimethamine and Amodiaquine (SPAQ) used in standard age-based dosing regimens for Seasonal Malaria Chemoprevention (SMC) in children 3-59 months and (2) determine the prevalences and associations of drug resistance genotypes associated with resistance to SPAQ.

1. a prospective cohort study to determine the chemoprevention efficacy of SPAQ (if SPAQ provides 28 days of protection from Plasmodium falciparum (P. falciparum) malaria infection by clearing existing and preventing new infections) and whether drug concentrations and/or resistance influence the ability to clear and prevent these P. falciparum infections.
2. a resistance markers study in symptomatic RDT positive children 3-59 months to measure sulfadoxine-pyrimethamine and amodiaquine resistance marker prevalence and association.

ELIGIBILITY:
Inclusion criteria

* Children between 3-59 months.
* Being resident in the research study area.
* Afebrile children with no other malaria associated symptoms in the past 48 hours or at time of recruitment.
* Consent to participate in the study obtained.
* Can comply with 3 days DOT of standard SPAQ regimen.
* Willingness and ability of the child's guardians to comply with the study protocol for the duration of the study including all dry blood spot and slide collections.

Exclusion criteria

* Symptoms of malaria (tympanic fever ≥ 37.5 °C or history of fever in past 48 hours)
* Known allergy to SPAQ.
* Receiving a sulfa-based medication for treatment or prophylaxis, including co-trimoxazole (trimethoprim-sulfamethoxazole).
* Individuals receiving azithromycin due to the antimalarial activity of azithromycin.
* Severe malnutrition according to WHO guidelines
* HIV positive or ARV use (SPAQ MUST NEVER be used with children taking the antiretroviral efavirenz)
* Chronic illness of any kind.
* Treatment with an ACT in previous 2 weeks.
* Previous treatment with SPAQ this malaria season.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Chemoprevention failure as defined by qPCR positive parasites or malaria slide positive parasites | 28 days
  Malaria slides and dry blood spots (DBS) taken at days 0,7,14, 21, 28 of a one month drug administration cycle will be analysed to detect parasitemia in children treated with SPAQ. Chemoprevention failure has occured if a malaria slide is positive for parasites 7 days or more after drug administration or if a qPCR detects low level parasitemia at the end of the administration cycle (one month).
Prevalence of antimalarial resistance markers among chemoprevention failures (as defined in outcome 1) | 28 days
  All Dried blood spots (DBS) will be analysed for malaria mutation genotypes (dhfr, dhps, Pfcrt, pfmdr1) on baseline and endline and additionally throughout the cycle if a chemoprevention failure (as defined in outcome 1) has occured.
Drug concentrations of Sulfadoxine-pyrimethamine and amodiaquine among chemoprevention failures (as defined in outcome 1) | 28 days
  Drug concentrations of SPAQ will be analyzed on all samples (taken at days 7,14,21,28 throughout the one month cycle) in order to be linked to chemoprevention failures as defined in outcome 1.
Prevalence over time of parasites with dhfr/dhps/pfcrt/pfmdr1 mutations in symptomatic children with a positive diagnostic test residing in districts where SMC is implemented | 28 days preceding implementation of chemoprevention efficacy study component
  The outcome measure to meet the secondary objective is the prevalence of molecular markers associated with SP (codons 108, 51 and 59 in dhfr and 437, 540 and 581 in dhps) and amodiaquine (codons 72-76 Pfcrt and 86, 184 and 1246 pfmdr1), as well as other markers of parasite genetic diversity, in blood samples collected from symptomatic children under five years with a positive RDT attending selected health facilities in areas with SMC

CONTACTS AND LOCATIONS:
Overall Officials: Craig Bonnington, Principal Investigator — Malaria Consortium
Locations (1):
- Kwara Sentinell Site, Kwara, Nigeria

IPD SHARING:
Plan to Share IPD: No